CLINICAL TRIAL: NCT07066163
Title: SMART-PD: Evaluating the Impact of Smartphone-Based Wearable Technology on Motor Symptoms and Quality of Life in People With Parkinson's Disease
Acronym: SMART PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other)
Responsible Party: Principal Investigator, Deepa Dash, Assistant Professor, Western University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 126861
Record Dates: First submitted 2025-06-05; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease, Idiopathic
Keywords: parkinson; wearable
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: video based assessment without knowledge of arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wearable device group (WDG): (Experimental): Participants who were randomized to the WDG will receive a smart watch and a mobile phone with KinesiaU application loaded. Participants will get hands on training on the first visit about how to use the smartwatch, how to enter medication details and access the reports on the phone. They will be instructed to wear the smartwatch for at least five out of seven days following the first visit.
  Interventions: Device: Kinesia U
- control group (Other): Participants in the control group will receive standard of care, consisting of regular management of their motor symptoms and monitoring using motor dairy, interview by their neurologist, family physician, and other healthcare providers. n.
  Interventions: Other: Standard of care treatment

INTERVENTIONS:
Device: Kinesia U — KinesiaU is a commercially available wearable technology, which includes a smart watch and a mobile application which can continuously monitor and quantify motor symptoms such as tremor, bradykinesia, dyskinesia, gait parameters throughout the day. The technology has been validated for motor symptoms and has high agreement with clinician ratings of motor severity. The motion sensor records data using KinesiaU smart watch and is then transmitted to a secure cloud database, where specialized algorithms analyze the information to detect motor symptoms and compute severity scores every 2 minutes. The results are then not only available to clinicians in the form of detailed reports for review but also for PwP in easily understandable format on the phone application . The validity of this device has been studied to assess tremor, bradykinesia and dyskinesia.
  Arms: Wearable device group (WDG):
Other: Standard of care treatment — Participants in the control group will receive standard of care, consisting of regular management of their motor symptoms and monitoring using motor dairy, interview by their neurologist, family physician, and other healthcare providers.
  Arms: control group

SUMMARY:
This study aims to evaluate whether wearable technology can improve the management of motor symptoms in people with Parkinson's disease (PD) who experience motor fluctuations throughout the day. The project will use a smartwatch and mobile app (KinesiaU) to continuously track movement, allowing for more responsive and personalized treatment compared to traditional monitoring methods.

In this pilot randomized controlled trial, 32 participants will be assigned to either:

A control group receiving standard care, or

A wearable device group receiving standard care plus using the smartwatch.

Outcomes will be assessed over a 4-week period, focusing on changes in motor function, quality of life, and self-management. The study will also examine feasibility, adherence, and data quality.

If successful, this trial will provide critical evidence for integrating wearable devices into routine clinical care for PD, paving the way for larger efficacy trials and more patient-centered care strategies.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common brain disorder that affects movement. It usually develops later in life and gradually worsens over time. People with Parkinson's may experience symptoms such as shaking (tremor), slow movement (bradykinesia), muscle stiffness, and problems with walking or balance. What makes Parkinson's especially challenging is that these symptoms can change throughout the day - a person may feel relatively well one moment and struggle to move just hours later.

Why is this a problem? This daily fluctuation in symptoms - known as motor fluctuations - makes it difficult for both patients and doctors to manage the disease. Traditional ways of monitoring symptoms, like keeping a diary or waiting until the next doctor's visit, don't always capture the full picture of what's happening. This can lead to treatment plans that don't match a person's actual needs.

What is the study about? We are exploring whether using wearable technology - in this case, a smartwatch and mobile app called KinesiaU - can help people with Parkinson's and their doctors better track and manage symptoms. The smartwatch measures movement throughout the day and sends data to a mobile app. This gives a more accurate and detailed view of how symptoms change over time, outside of the doctor's office.

Who is involved in the study?

The study will include 32 people living with Parkinson's disease who are experiencing motor fluctuations. They will be randomly divided into two groups:

Group 1: Standard Care Group - These participants will continue their regular care, which may include doctor visits, motor symptom diaries, and interviews with their care team.

Group 2: Wearable Device Group - These participants will also receive standard care plus use the KinesiaU smartwatch and app. They will wear the device at least five days a week, and the information it collects will be used by their doctors to make timely and personalized treatment decisions.

How will the study work?

Everyone in the study will be assessed at the beginning, then again at Week 2 and Week 4. During these check-ins,Investigators will measure:

Changes in movement symptoms using a standard clinical scale (MDS-UPDRS III)

Quality of life (using a questionnaire called PDQ-39)

How confident patients feel in managing their health (using a tool called PAM-13)

Investigators will also track whether people are willing and able to stick with the program, how often they wear the device, and whether the data collected is complete and usable.

Why is this study important? This is the first pilot study in our region to test this kind of wearable technology for people with Parkinson's. If it goes well, it will show that using a smartwatch is not only possible and helpful, but also something people are willing to do. The results will guide a larger study in the future and could help bring this kind of technology into routine clinical care.

The goal is to make Parkinson's care more personalized, data-driven, and responsive to real life. Investigators believe that by using innovative tools like smartwatches, we can give people living with Parkinson's more control over their health and improve their quality of life.

ELIGIBILITY:
Inclusion criteria:

* Meet criteria for Parkinson's disease using MDS Clinical Diagnostic Criteria for Parkinson's Disease
* Presence of Motor fluctuations based on movement disorder neurologist assessment.
* Motor ability to use the wearable device and access the wearable device application.
* Cognitively ability to do ADL's and use the wearable device and access the wearable device application based on clinician's judgment.
* Knowledge of English to enter medication details in the wearable device application.

Exclusion criteria:

* Physical barriers in using the wearable device.
* Atypical Parkinsonian disorder or other causes of Parkinsonism
* Inability to read or write English.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Through study completion, an average of 1 year".
  Recruitment rate, defined as the number of participants recruited divided by the number of participants eligible, multiplied by 100. This will indicate how effectively the study was able to enroll suitable participants.
Retention Rate | Through study completion, around 1year
  Retention rate calculated as the number of participants who complete the study divided by those recruited, and the dropout rate as the number of participan
Completion of Intervention: | Through study completion, around 1year
  The proportion of participants adhering to the full intervention will be calculated

SECONDARY OUTCOMES:
MDS Unified Parkinson's Disease Rating Scale Part 3 | 4 weeks
  MDS UPDRS is a validated tool specifically used to assess motor severity in PwP. It measures a range of motor symptoms, including tremor, rigidity, bradykinesia, and postural instability, providing a comprehensive evaluation of motor impairment.

OTHER OUTCOMES:
Therapy Adjustments | 4 weeks
  * Change in medication from baseline to week 4 to capture increase or decrease in dosage, change in medications, adding new medications
  * Change in advanced therapeutic interventions from baseline to week 4 to capture changes in deep brain stimulation parameters or referral for advanced therapies
Quality of life | 4 WEEKS
  Change in Parkinson's Disease Questionnaire-39 (PDQ-39) score is a validated patient- reported outcome measure widely used in clinical trials and research to assess the quality of life in individuals with Parkinson's disease (PD). It evaluates the impact of PD on daily life across 8 domains and has 39 questions. Each item is scored on a 5-point Likert scale, where 0 = Never, 1 = Occasionally, 2 = Sometimes, 3 = Often, and 4 = Always. The scores for each domain are transformed into a scale of 0 to 100, with higher scores indicating worse health and quality of life.
Adverse events | 4 weeks
  Adverse events realted to the use of the smart watch

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - London Health Sciences Center.London ,Ontario, London, Ontario
  - London Health Sciences Center, London, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
As a small-scale feasibility study involving only 32 participants, the dataset may not be robust enough to support secondary analyses or generalizable conclusions. Sharing such limited data could risk misinterpretation or misuse.